CLINICAL TRIAL: NCT03791775
Title: A Multicentre, Open-label, Single-arm Phase II Trial on the Efficacy and Safety of Sclerotherapy Using 3% Polidocanol Foam to Treat Second-degree Hemorrhoidal Disease
Brief Title: Efficacy and Safety of Polidocanol Foam 3% in the Treatment of II Degree Hemorrhoidal Disease
Acronym: SCLEROFOAM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Collaborators: SICCR - Gaetano Gallo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 274/2018
Record Dates: First submitted 2018-12-29; First posted 2019-01-03 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Second-degree Hemorrhoids
Keywords: Hemorrhoids; Sclerotherapy; Polidocanol 3%; Non-surgical treatments
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study, according to the inclusion and exclusion criteria, will undergo sclerotherapy performed with polidocanol foam (Atossisclerol® 3%, Chemische Fabrik Kreussler & Co. GmbH, Wiesbaden, Germany).
  The procedure will be performed in the Sims position or lithotomy position. A modified Blonde-Blanchard technique will be adopted, with the tangential injection of polidocanol foam into the submucosa of the apex of each hemorrhoidal pile, without exceeding three piles, and using a self-lighting open-ended anoscope and a 20-G needle in order to reduce bleeding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polidocanol 3% Foam (Experimental): Patients enrolled in the study, according to the inclusion and exclusion criteria, will undergo sclerotherapy performed with polidocanol foam (Atossisclerol® 3%, Chemische Fabrik Kreussler & Co. GmbH, Wiesbaden, Germany).
  Interventions: Drug: Polidocanol foam (Atossisclerol® 3%)

INTERVENTIONS:
Drug: Polidocanol foam (Atossisclerol® 3%) — The procedure will be performed in the Sims position or lithotomy position. A modified Blonde-Blanchard technique will be adopted, with the tangential injection of polidocanol foam into the submucosa of the apex of each hemorrhoidal pile, without exceeding three piles, and using a self-lighting open-ended anoscope and a 20-G needle in order to reduce bleeding

SUMMARY:
Hemorrhoidal disease (HD) is one of the oldest and most common proctologic diseases that has been described with an estimated prevalence between 4.4% and 86%. Despite the proposal of three mechanisms that might underlie haemorrhoidal development - the varicose vein theory, the vascular hyperplasia theory and the sliding anal-lining theory, the exact pathophysiology of symptomatic hemorrhoid disease is poorly understood.

HD seems to be the most common cause for rectal bleeding, or hematochezia, and the second most frequent cause for severe rectorrhagia after diverticulitis. The blood is bright red and coats the stool at the end of defection. Other symptoms include pain, mucous discharge, itching or the sensation of tissue prolapse.

The most widely accepted classification is the Goligher classification:

* Grade I: hemorrhoids bleed but do not prolapse out of the anal canal;
* Grade II: hemorrhoidal cushions prolapse outside of the anal canal on straining or during bowel movements, but reduce spontaneously;
* Grade III: hemorrhoidal cushions prolapse outside the anal canal on straining and require manual reduction;
* Grade IV: hemorrhoidal prolapse is irreducible even with manipulation

DETAILED DESCRIPTION:
As reported by the guidelines of the Italian Society of Colorectal Surgery, in case of failure of conservative therapies the most common outpatient treatments for first- and second-degree Hemorrhoidal Disease (HD) are rubber band ligation and sclerotherapy.

Sclerotherapy causes an inflammatory reaction with local sclerosis of the submucosal tissue and a consequent fixation of the haemorrhoidal tissue to the underlying tissue. Moreover, the effect of sclerosing solutions is that of making vascular damage via producing endothelial injury.

A 100% improvement in bleeding was reported in patients with II and grade III hemorrhoids, and a complete resolution of the condition was described in 69% of non-selected patients, 52% in grade III and 88% in grade I. Resolution of prolapse was reported in 90-100% of patients affected by grade II hemorrhoids. Complications are rare but serious, and include impotence, irreversible necrotizing fasciitis and abdominal compartment syndrome [31-33]. In Germany, sclerotherapy with liquid agents is considered the first choice in treating grade I hemorrhoids. The only approved medical product by German authorities is polidocanol (Lauromacrogol 400 (INN), H3C-(CH2)11-(O-CH2-CH2)n∼9-OH), produced by Chemische Fabrik Kreussler & Co. GmbH.

In Italy, this drug is known as Atossisclerol 3%. The polidocanol is a non-ionic detergent made up of a chain of hydrophilic polyethylene oxide mixed with aliphatic hydrophobic dodecyl alcohol and it is recommended for first- and second-degree HD. The effects of polidocanol are similar to those of phenol oil but less number of side effects.

Based on these experiences, Karl-Heinz Moser introduced the use of polidocanol foam in the treatment of grade I hemorrhoids. In 2013, the same author published the results of a randomized, controlled, single blind, multicentre trial on the efficacy and safety of sclerotherapy with polidocanol foam in comparison with liquid sclerosant agents in treating grade I hemorrhoids [28]. In the foam group success rate after one sclerotherapy session was 88%, while success rate among patients treated with liquid polidocanol was 69%. Furthermore, patients treated with foam were more satisfied than those treated with liquid polidocanol (99% vs. 84% p=0.009). Finally, the quantity of polidocanol injected in the foam group was significantly lower (p<0.001), as well as the number of sessions requested (p<0.001).

In summary, according to the authors, these results suggest that polidocanol foam can be used as the treatment of choice in grade I HD.

The aim of this study is to evaluate the efficacy and safety of sclerotherapy with 3% polidocanol foam (PF) on patients affected by second-degree HD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 18 and below 75 years of age with a confirmed diagnosis of second-degree HD (proctological examination, proctoscopy and, if required, colonoscopy)
2. Patients who report persistent perianal bleeding as a typical symptom of second-degree HD
3. Informed consent from each patient must be obtained
4. Participating centres will be asked to confirm that they have gained formal approval at their site

Exclusion Criteria:

1. Previous anal surgical procedures
2. Previous sclerotherapy or rubber band ligation in the last 12 months
3. Positive pregnancy test
4. Patients with inability to return for postoperative control visits, to sign the informed consent or to fill out the required clinical diary
5. Breast-feeding
6. Known allergy to polidocanol
7. Acute perianal thrombosis
8. Anal fistula
9. Anal fissure
10. Proctitis
11. Fecal incontinence
12. Coagulation disorders
13. Anticoagulant therapy
14. Known HBV, HCV and HIV infection
15. Acite Crohn's disease or Ulcerative colitis
16. Diabetes mellitus I and II
17. COPD
18. Any kind of tumour
19. Previous pelvic radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Success Rate 1 | 12 months follow-up
  To establish the success rate after one sclerotherapy session, in terms of complete resolution of bleeding episodes one week after the injection
  Bleeding will be assessed using both the Hemorrhoidal Disease Symptoms Score and the Giamundo score.
  Rørvik HD et al (2019) Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum; 62:333-342
  Giamundo et al (2018) Doppler-guided hemorrhoidal dearterialization with laser (HeLP): a prospective analysis of data from a multicenter trial. Tech Coloproctol; 25:635-643

SECONDARY OUTCOMES:
Success Rate 2 | 12 months follow-up
  To establish the success rate in terms of partial or complete resolution of the symptoms
  Symptoms will be assessed using the Hemorrhoidal Disease Symptom Score described by Rorvik HD
Number of outpatient sessions | 12 months follow-up
  To evaluate the average number of outpatient sessions necessary for treatment success
Rate of complications - adverse events | 6 months follow-up
  To establish the rate of complications
Quality of Life | 12 months follow-up
  Short Health Scale HD
  4 questions with 7-point Liker scale each (1 = very dissatisfied, 7 = very satisfied)
  Minimum = 4
  Maximum = 28
To establish the average time required to reach autonomy | 12 months follow-up
  We considered autonomy as the return to normal activity: it includes also the return to work apart from cases of retired patients in which we considered it as the complete return to daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Gallo, MD, Principal Investigator — Department of Medical and Surgical Sciences, University of Catanzaro, Catanzaro 88100, Italy
Locations (1):
- University of Catanzaro, Catanzaro, Italy

REFERENCES:
- [Background] Akerud L (1995) Sclerotherapy of haemorrhoids: a prospective randomised trial of polidocanol and phenol in oil. Coloproctology 17:73-86
- [Background] Moser KH (2007) Evaluation of the efficacy and safety of polidocanol foam in the sclerotherapy of first degree bleeding haemorrhoids. Phlebol Rev (Przeglad Flebologiczny) 15:103-106
- [Background] Blanchard CE (1928) Textbook of ambulant proctology p. 134. Medical Success Press, Youngstown Ohio
- [Background] Gallo G, Sacco R, Sammarco G (2018) Epidemiology of Hemorrhoidal Disease. In: Hemorrhoids. Coloproctology (eds Ratto C, Parello A, Litta F), vol 2. Cham: Springer pp. 3-7
- [Result] Thomson WH. The nature of haemorrhoids. Br J Surg. 1975 Jul;62(7):542-52. doi: 10.1002/bjs.1800620710. PMID 1174785
- [Result] Aigner F, Bodner G, Gruber H, Conrad F, Fritsch H, Margreiter R, Bonatti H. The vascular nature of hemorrhoids. J Gastrointest Surg. 2006 Jul-Aug;10(7):1044-50. doi: 10.1016/j.gassur.2005.12.004. PMID 16843876
- [Result] Burkitt DP. Varicose veins, deep vein thrombosis, and haemorrhoids: epidemiology and suggested aetiology. Br Med J. 1972 Jun 3;2(5813):556-61. doi: 10.1136/bmj.2.5813.556. PMID 5032782
- [Result] Gralnek IM, Ron-Tal Fisher O, Holub JL, Eisen GM. The role of colonoscopy in evaluating hematochezia: a population-based study in a large consortium of endoscopy practices. Gastrointest Endosc. 2013 Mar;77(3):410-8. doi: 10.1016/j.gie.2012.10.025. Epub 2013 Jan 5. PMID 23294756
- [Result] Nikpour S, Ali Asgari A. Colonoscopic evaluation of minimal rectal bleeding in average-risk patients for colorectal cancer. World J Gastroenterol. 2008 Nov 14;14(42):6536-40. doi: 10.3748/wjg.14.6536. PMID 19030208
- [Result] Wong RF, Khosla R, Moore JH, Kuwada SK. Consider colonoscopy for young patients with hematochezia. J Fam Pract. 2004 Nov;53(11):879-84. PMID 15527724
- [Result] Mehanna D, Platell C. Investigating chronic, bright red, rectal bleeding. ANZ J Surg. 2001 Dec;71(12):720-2. doi: 10.1046/j.1445-1433.2001.02277.x. PMID 11906386
- [Result] Gayer C, Chino A, Lucas C, Tokioka S, Yamasaki T, Edelman DA, Sugawa C. Acute lower gastrointestinal bleeding in 1,112 patients admitted to an urban emergency medical center. Surgery. 2009 Oct;146(4):600-6; discussion 606-7. doi: 10.1016/j.surg.2009.06.055. PMID 19789018
- [Result] Newman J, Fitzgerald JE, Gupta S, von Roon AC, Sigurdsson HH, Allen-Mersh TG. Outcome predictors in acute surgical admissions for lower gastrointestinal bleeding. Colorectal Dis. 2012 Aug;14(8):1020-6. doi: 10.1111/j.1463-1318.2011.02824.x. PMID 21910819
- [Result] Goligher JC. Cryosurgery for hemorrhoids. Dis Colon Rectum. 1976 Apr;19(3):213-8. doi: 10.1007/BF02590905. No abstract available. PMID 1269347
- [Result] Trompetto M, Clerico G, Cocorullo GF, Giordano P, Marino F, Martellucci J, Milito G, Mistrangelo M, Ratto C. Erratum to: Evaluation and management of hemorrhoids: Italian society of colorectal surgery (SICCR) consensus statement. Tech Coloproctol. 2016 Mar;20(3):201. doi: 10.1007/s10151-015-1416-0. No abstract available. PMID 26728606
- [Result] Awad AE, Soliman HH, Saif SA, Darwish AM, Mosaad S, Elfert AA. A prospective randomised comparative study of endoscopic band ligation versus injection sclerotherapy of bleeding internal haemorrhoids in patients with liver cirrhosis. Arab J Gastroenterol. 2012 Jun;13(2):77-81. doi: 10.1016/j.ajg.2012.03.008. Epub 2012 Apr 24. PMID 22980596
- [Result] Forlini A, Manzelli A, Quaresima S, Forlini M. Long-term result after rubber band ligation for haemorrhoids. Int J Colorectal Dis. 2009 Sep;24(9):1007-10. doi: 10.1007/s00384-009-0698-y. Epub 2009 Apr 23. PMID 19387663
- [Result] Kanellos I, Goulimaris I, Christoforidis E, Kelpis T, Betsis D. A comparison of the simultaneous application of sclerotherapy and rubber band ligation, with sclerotherapy and rubber band ligation applied separately, for the treatment of haemorrhoids: a prospective randomized trial. Colorectal Dis. 2003 Mar;5(2):133-8. doi: 10.1046/j.1463-1318.2003.00395.x. PMID 12780901
- [Result] Fukuda A, Kajiyama T, Arakawa H, Kishimoto H, Someda H, Sakai M, Tsunekawa S, Chiba T. Retroflexed endoscopic multiple band ligation of symptomatic internal hemorrhoids. Gastrointest Endosc. 2004 Mar;59(3):380-4. doi: 10.1016/s0016-5107(03)02818-9. PMID 14997135
- [Result] Bernal JC, Enguix M, Lopez Garcia J, Garcia Romero J, Trullenque Peris R. Rubber-band ligation for hemorrhoids in a colorectal unit. A prospective study. Rev Esp Enferm Dig. 2005 Jan;97(1):38-45. doi: 10.4321/s1130-01082005000100005. English, Spanish. PMID 15801896
- [Result] Gupta PJ, Heda PS, Kalaskar S. Randomized controlled study between suture ligation and radio wave ablation and suture ligation of grade III symptomatic hemorrhoidal disease. Int J Colorectal Dis. 2009 Apr;24(4):455-60. doi: 10.1007/s00384-008-0579-9. Epub 2008 Sep 7. PMID 18777127
- [Result] Iyer VS, Shrier I, Gordon PH. Long-term outcome of rubber band ligation for symptomatic primary and recurrent internal hemorrhoids. Dis Colon Rectum. 2004 Aug;47(8):1364-70. doi: 10.1007/s10350-004-0591-2. PMID 15484351
- [Result] Wehrmann T, Riphaus A, Feinstein J, Stergiou N. Hemorrhoidal elastic band ligation with flexible videoendoscopes: a prospective, randomized comparison with the conventional technique that uses rigid proctoscopes. Gastrointest Endosc. 2004 Aug;60(2):191-5. doi: 10.1016/s0016-5107(04)01551-2. PMID 15278043
- [Result] Beattie GC, Rao MM, Campbell WJ. Secondary haemorrhage after rubber band ligation of haemorrhoids in patients taking clopidogrel--a cautionary note. Ulster Med J. 2004 Nov;73(2):139-41. No abstract available. PMID 15651778
- [Result] Chau NG, Bhatia S, Raman M. Pylephlebitis and pyogenic liver abscesses: a complication of hemorrhoidal banding. Can J Gastroenterol. 2007 Sep;21(9):601-3. doi: 10.1155/2007/106946. PMID 17853956
- [Result] Tejirian T, Abbas MA. Bacterial endocarditis following rubber band ligation in a patient with a ventricular septal defect: report of a case and guideline analysis. Dis Colon Rectum. 2006 Dec;49(12):1931-3. doi: 10.1007/s10350-006-0769-x. PMID 17080276
- [Result] Sim HL, Tan KY, Poon PL, Cheng A, Mak K. Life-threatening perineal sepsis after rubber band ligation of haemorrhoids. Tech Coloproctol. 2009 Jun;13(2):161-4. doi: 10.1007/s10151-008-0435-5. Epub 2008 Aug 5. PMID 18679564
- [Result] Yano T, Asano M, Tanaka S, Oda N, Matsuda Y. Prospective study comparing the new sclerotherapy and hemorrhoidectomy in terms of therapeutic outcomes at 4 years after the treatment. Surg Today. 2014 Mar;44(3):449-53. doi: 10.1007/s00595-013-0564-y. Epub 2013 Mar 30. PMID 23543083
- [Result] Miyamoto H, Asanoma M, Miyamoto H, Shimada M. ALTA injection sclerosing therapy:non-excisional treatment of internal hemorrhoids. Hepatogastroenterology. 2012 Jan-Feb;59(113):77-80. doi: 10.5754/hge11089. PMID 22260824
- [Result] Tokunaga Y, Sasaki H. Impact of less invasive treatments including sclerotherapy with a new agent and hemorrhoidopexy for prolapsing internal hemorrhoids. Int Surg. 2013 Jul-Sep;98(3):210-3. doi: 10.9738/INTSURG-D-13-00030.1. PMID 23971772
- [Result] Moser KH, Mosch C, Walgenbach M, Bussen DG, Kirsch J, Joos AK, Gliem P, Sauerland S. Efficacy and safety of sclerotherapy with polidocanol foam in comparison with fluid sclerosant in the treatment of first-grade haemorrhoidal disease: a randomised, controlled, single-blind, multicentre trial. Int J Colorectal Dis. 2013 Oct;28(10):1439-47. doi: 10.1007/s00384-013-1729-2. Epub 2013 Jun 18. PMID 23775099
- [Result] Takano M, Iwadare J, Ohba H, Takamura H, Masuda Y, Matsuo K, Kanai T, Ieda H, Hattori Y, Kurata S, Koganezawa S, Hamano K, Tsuchiya S. Sclerosing therapy of internal hemorrhoids with a novel sclerosing agent. Comparison with ligation and excision. Int J Colorectal Dis. 2006 Jan;21(1):44-51. doi: 10.1007/s00384-005-0771-0. Epub 2005 Apr 21. PMID 15843937
- [Result] Yano T, Nogaki T, Asano M, Tanaka S, Kawakami K, Matsuda Y. Outcomes of case-matched injection sclerotherapy with a new agent for hemorrhoids in patients treated with or without blood thinners. Surg Today. 2013 Aug;43(8):854-8. doi: 10.1007/s00595-012-0365-8. Epub 2012 Oct 10. PMID 23052752
- [Result] Bullock N. Impotence after sclerotherapy of haemorrhoids: case reports. BMJ. 1997 Feb 8;314(7078):419. doi: 10.1136/bmj.314.7078.419. No abstract available. PMID 9040388
- [Result] Schulte T, Fandrich F, Kahlke V. Life-threatening rectal necrosis after injection sclerotherapy for haemorrhoids. Int J Colorectal Dis. 2008 Jul;23(7):725-6. doi: 10.1007/s00384-007-0402-z. Epub 2007 Nov 28. No abstract available. PMID 18043926
- [Result] Yang P, Wang YJ, Li F, Sun JB. Hemorrhoid sclerotherapy with the complication of abdominal compartment syndrome: report of a case. Chin Med J (Engl). 2011 Jun;124(12):1919-20. PMID 21740855
- [Result] Lobascio P, Minafra M, Laforgia R, Giove C, Trompetto M, Gallo G. The use of sclerotherapy with polidocanol foam in the treatment of second-degree haemorrhoidal disease - a video vignette. Colorectal Dis. 2019 Feb;21(2):244-245. doi: 10.1111/codi.14498. Epub 2018 Dec 15. No abstract available. PMID 30485654
- [Result] Namasivayam J, Payne D, Maguire D. Prostatic abscess following injection of internal haemorrhoids. Clin Radiol. 2000 Jan;55(1):67-8. doi: 10.1053/crad.1999.0066. No abstract available. PMID 10650114
- [Result] Barwell J, Watkins RM, Lloyd-Davies E, Wilkins DC. Life-threatening retroperitoneal sepsis after hemorrhoid injection sclerotherapy: report of a case. Dis Colon Rectum. 1999 Mar;42(3):421-3. doi: 10.1007/BF02236364. PMID 10223767
- [Result] Kaman L, Aggarwal S, Kumar R, Behera A, Katariya RN. Necrotizing fascitis after injection sclerotherapy for hemorrhoids: report of a case. Dis Colon Rectum. 1999 Mar;42(3):419-20. doi: 10.1007/BF02236363. PMID 10223766
- [Result] Wollmann JC. The history of sclerosing foams. Dermatol Surg. 2004 May;30(5):694-703; discussion 703. doi: 10.1111/j.1524-4725.2004.30208.x. PMID 15099310
- [Result] Yamaki T, Nozaki M, Iwasaka S. Comparative study of duplex-guided foam sclerotherapy and duplex-guided liquid sclerotherapy for the treatment of superficial venous insufficiency. Dermatol Surg. 2004 May;30(5):718-22; discussion 722. doi: 10.1111/j.1524-4725.2004.30202.x. PMID 15099313
- [Result] Rabe E, Otto J, Schliephake D, Pannier F. Efficacy and safety of great saphenous vein sclerotherapy using standardised polidocanol foam (ESAF): a randomised controlled multicentre clinical trial. Eur J Vasc Endovasc Surg. 2008 Feb;35(2):238-45. doi: 10.1016/j.ejvs.2007.09.006. Epub 2007 Nov 7. PMID 17988905
- [Result] Ouvry P, Allaert FA, Desnos P, Hamel-Desnos C. Efficacy of polidocanol foam versus liquid in sclerotherapy of the great saphenous vein: a multicentre randomised controlled trial with a 2-year follow-up. Eur J Vasc Endovasc Surg. 2008 Sep;36(3):366-70. doi: 10.1016/j.ejvs.2008.04.010. Epub 2008 Jun 3. PMID 18524643
- [Result] BARRON J. Office ligation of internal hemorrhoids. Am J Surg. 1963 Apr;105:563-70. doi: 10.1016/0002-9610(63)90332-5. No abstract available. PMID 13969563
- [Result] Rorvik HD, Styr K, Ilum L, McKinstry GL, Dragesund T, Campos AH, Brandstrup B, Olaison G. Hemorrhoidal Disease Symptom Score and Short Health ScaleHD: New Tools to Evaluate Symptoms and Health-Related Quality of Life in Hemorrhoidal Disease. Dis Colon Rectum. 2019 Mar;62(3):333-342. doi: 10.1097/DCR.0000000000001234. PMID 30451751
- [Result] Giamundo P, Braini A, Calabro' G, Crea N, De Nardi P, Fabiano F, Lippa M, Mastromarino A, Tamburini AM. Doppler-guided hemorrhoidal dearterialization with laser (HeLP): a prospective analysis of data from a multicenter trial. Tech Coloproctol. 2018 Aug;22(8):635-643. doi: 10.1007/s10151-018-1839-5. Epub 2018 Aug 29. PMID 30159627